CLINICAL TRIAL: NCT05325138
Title: Assessing Knowledge, Beliefs and Attitudes Toward HPV Vaccination Among Parents With Children Aged 9-14yrs Within Rural Communities in North West Region, Cameroon
Brief Title: Assessing Knowledge, Beliefs and Attitudes Toward HPV Vaccination Among Parents in North West, Cameroon
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Principal Investigator, Lorraine Elit, MD, Professor Emeritus, McMaster University
Other Study IDs: 100035
Record Dates: First submitted 2022-01-10; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Vaccine Refusal
Keywords: HPV vaccine, parental perspective, qualitative study
MeSH Terms: conditions — Vaccination Refusal | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parents: Parents of girls aged 9-14 years old
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Parents of girls aged 9-14yearsold will undergo an interview to determine their knowledge, attitudes and beliefs concerning HPV vaccination

SUMMARY:
The aim of this study is to assess knowledge, beliefs and attitudes of parents to young girls aged 9 to 14 years about HPV vaccines within some rural communities in the North West Region of Cameroon served by three hospitals in that area. To do this, we will conduct in-depth qualitative interviews with purposively sampled parents of girls aged 9 to 14 years, some of whom received HPV vaccine and some of whom did not. Interviews will continue until thematic saturation is reached (We anticipate a total 40 interviews). Data analysis will be done concurrently with interviews using thematic analysis.

DETAILED DESCRIPTION:
The aim of this study is to assess knowledge, beliefs and attitudes of parents to young girls aged 9 to 14 years about HPV vaccines within some rural communities in the North West Region of Cameroon served by three hospitals in that area. Snowball sampling technique will be used. Parents of girls aged 9-14years will be included if the daughters have or have not received the HPV vaccine. Exclusion criteria include parents who are health care workers in any health institution, unwilling to provide consent, or inability to converse in English or pidgeon English. In-depth one-on-one interviews will take place using an interview guide. Interviews will be in English or pidgeon English. They will be taped and transcribed. Data will be entered into ATLAS Ti. Data analysis will be done concurrently with interviews using thematic analysis.Interviews will continue until theme saturation is reached (We anticipate a total 40 interviews).

ELIGIBILITY:
Inclusion Criteria:

* Parents of girls aged 9-14 years old living in Mbingo, Njinikom or Fundong health areas of northwestern Cameroon.

Exclusion Criteria:

* Parents who are health care workers or working in any health institution.
* Not willing to provide informed consent
* Not able to converse in English or pidgeon English

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents of girls aged 9-14 years old living in rural north western Cameroon (Mbingo, Njinikom, or Fundong). Their daughters may or may not have received the HPV vaccine.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
HPV vaccine knowledge, attitudes and beliefs | 6months
  Interviews of parents of girls (ages 9-14 years old)

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine M Elit, MD MSc, Principal Investigator — McMaster University
Locations (1):
- Mbingo Hosptial, Bamenda, North-West Region, Cameroon

IPD SHARING:
Plan to Share IPD: No
No IPD sharing is planned

REFERENCES:
- [Derived] Elit L, Tum EM, Ngalla C, Fungchwi GM, Fokom Domgue J, Nouvet E. Perceptions of Cancer in Parents of Adolescent Daughters in Northwest Cameroon. Curr Oncol. 2023 Jul 25;30(8):7167-7177. doi: 10.3390/curroncol30080519. PMID 37623000
- [Derived] Elit L, Ngalla C, Afugchwi GM, Tum E, Fokom Domgue J, Nouvet E. Assessing knowledge, attitudes and belief toward HPV vaccination of parents with children aged 9-14 years in rural communities of Northwest Cameroon: a qualitative study. BMJ Open. 2022 Nov 15;12(11):e068212. doi: 10.1136/bmjopen-2022-068212. PMID 36379650
- [Derived] Elit L, Ngalla C, Afugchwi GM, Tum E, Fokom-Domgue J, Nouvet E. Study protocol for assessing knowledge, attitudes and belief towards HPV vaccination of parents with children aged 9-14 years in rural communities of North West Cameroon: a qualitative study. BMJ Open. 2022 Aug 24;12(8):e062556. doi: 10.1136/bmjopen-2022-062556. PMID 36002223